CLINICAL TRIAL: NCT00281242
Title: Innate and Adaptive Immunity in COPD Exacerbations: Severe AE-COPD Clinical Course Study
Brief Title: Changes in Cytokine Levels During an Acute Exacerbation of Chronic Obstructive Pulmonary Disease
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Jeffrey L. Curtis, Professor of Internal Medicine (Pulmonary & Critical Care Medicine), University of Michigan
Other Study IDs: 1325; R01HL082480 (NIH)
Record Dates: First submitted 2006-01-20; First posted 2006-01-24 (Estimated); Last update posted 2016-01-29 (Estimated); Status verified 2016-01

CONDITIONS: Pulmonary Disease, Chronic Obstructive; Lung Diseases, Obstructive
Keywords: Chronic Obstructive Pulmonary Disease; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Lung Diseases, Obstructive | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Research subjects: All participants undergo the same testing in this observational trial. There is no randomization, and no interventions other than blood drawing.
  Interventions: Other: blood draw

INTERVENTIONS:
Other: blood draw — All subjects undergo blood draws at study visits and at the time of COPD exacerbation visits.

SUMMARY:
The purpose of this study is to determine whether there is a statistical association between changes in sputum serial levels of two cytokines, interleukin (IL)-17 and IL-6, during the treatment course of a severe acute exacerbation of chronic obstructive pulmonary disease (AE-COPD) and during the clinical course itself (i.e., rate of recovery or potential complicated course). AE-COPD is defined as an episode requiring emergency room (ER) evaluation.

DETAILED DESCRIPTION:
BACKGROUND:

COPD is one of the most pressing healthcare problems facing our nation. AE-COPD is responsible for the bulk of healthcare costs, and much of the morbidity and decline in health status among individuals with this common disease. The lack of accepted animal models of AE-COPD necessitates novel approaches using human samples. Advances in the understanding of the pathogenesis have been slowed, in part, due to controversy as to how exacerbations should be defined. The prevailing paradigm has defined AE-COPD as event-based. Such definitions clearly identify groups of patients with accelerated loss of pulmonary function and increased mortality. However, limited data show that symptom-based definitions of AE-COPD also capture episodes inducing significant morbidity and functional decline, and hence of concern to patients. Fundamental mechanisms are lacking to explain AE-COPD defined by either means.

Controversy also surrounds triggers of AE-COPD. Bacteria and viruses are involved in some episodes, but the relative importance of each is intertwined with disputes over the definition of AE-COPD. Progress at linking specific pathogens to molecular pathogenesis has been slow, both due to their diversity, and to the high rates of bacterial colonization of patients with COPD, even in the stable state. Moreover, in many AE-COPD cases, no pathogen can be identified. Without negating the value of analyzing infections with specific species of pathogens, it appears that progress in molecular pathogenesis could be accelerated by focusing on unifying features of the pulmonary immune response during AE-COPD.

DESIGN NARRATIVE:

The research protocol will involve a prospective, observational analysis. Participants will include acutely ill COPD patients having an AE-COPD who are enrolled during an ER evaluation or hospitalization at Ann Arbor VA Hospital or the University of Michigan Health Systems ER, clinic, or wards. All non-study diagnostic testing, decisions to discharge from the ER or admit to hospital, prescription of medications, and non-study follow-up will be left to the discretion of the primary caregivers.

Participants who are either being or anticipate being discharged to their usual residence from the ER will be enrolled while still in the ER. Participants who were discharged to their usual residence may be contacted by telephone and enrolled up to 24 hours later, if willing to return to the Medical Center for study initiation. Hospitalized patients will be enrolled within the first 48 hours. Study physicians and coordinators will be on call to capture people at presentation, prior to steroids and antibiotics, if possible. However, clinically indicated treatment will not be delayed to permit enrollment or collection of research samples. Participants will be questioned about the status of five respiratory symptoms (dyspnea, cough, sputum production, sputum viscosity, sputum purulence) using a published Respiratory Symptom score instrument. Each symptom will be scored for severity using the following three-point scale: 1) Usual level; 2) Somewhat worse than usual; 3) Much worse than usual. An acute exacerbation of chronic bronchitis (AECB) will be defined symptomatically as a minor worsening (score of 2) for two or more symptoms, or a major worsening (score of 3) for one or more symptoms.

A clinical score will be generated using a previously used system (Chest 2000; 118:1557-1565) in which 10 clinical parameters will be assessed (overall feeling of well-being, dyspnea, cough, sputum production, sputum viscosity, sputum purulence, overall appearance, respiratory rate, wheezing, and rales); severity of each parameter will be scored using the same three-point scale. Thus the scores will range from 10 to 30.

The following additional data will be obtained: vital signs (blood pressure, pulse, temperature, respiratory rate, oxygen saturation level); dyspnea assessment (MMRC & University of California San Diego SOBQ); estimate of daily sputum production over last 72 hours; sputum color (using a standardized color "paint-chip" scale); changes in medication usage, with special attention to elicit any history of increased use of potent inhaled steroids, or patient-initiated use of oral steroids or antibiotics. If there is fever or focal findings on chest examination, a chest X-ray will be obtained as part of usual clinical care.

Sputum and blood samples will be collected for measurement of IL-6 and IL-17 levels at time 0 in the ER or hospital, and then 5-7 days, 10-12 days, 33-35 days, and 56-58 days later. Specimens may be obtained from participants requiring mechanical ventilation during the first 24 hours of intubation only, and only if they are not suspected to have pneumonia.

Subjects are reimbursed $25 per scheduled return visit following hospital discharge to help defray travel expenses.

ELIGIBILITY:
Inclusion criteria:

* Diagnosis of COPD (following American Thoracic Society guidelines) and/or chronic bronchitis
* ER visit and/or hospitalization with AE-COPD
* Current or former smokers with more than 20 pack-years
* Willingness to participate in follow-up studies defined in the protocol
* Ability to give informed consent

Exclusion criteria:

* Unstable cardiovascular disease
* Other systemic disease in which survival of more than 2 years is unlikely
* Mental incompetence or active psychiatric illness
* Currently taking more than 20 mg/day of Prednisone
* Participation in another experimental protocol within 6 weeks of study entry
* Asthma
* Cystic fibrosis
* Clinically significant bronchiectasis
* Lung cancer
* Other inflammatory or fibrotic lung disease

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Emergency room and clinics
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2005-09; Primary Completion 2010-06 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
biomarker analysis at the time of exacerbation, no clinical outcome | at each exacerbation

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey L. Curtis, Study Chair — University of Michigan at Ann Arbor
Locations (1):
- University of Michigan at Ann Arbor, Ann Arbor, Michigan, United States

REFERENCES:
- [Background] Curtis JL, Freeman CM, Hogg JC. The immunopathogenesis of chronic obstructive pulmonary disease: insights from recent research. Proc Am Thorac Soc. 2007 Oct 1;4(7):512-21. doi: 10.1513/pats.200701-002FM. PMID 17878463
- [Result] Freeman CM, Curtis JL, Chensue SW. CC chemokine receptor 5 and CXC chemokine receptor 6 expression by lung CD8+ cells correlates with chronic obstructive pulmonary disease severity. Am J Pathol. 2007 Sep;171(3):767-76. doi: 10.2353/ajpath.2007.061177. Epub 2007 Jul 19. PMID 17640964
- [Result] Freeman CM, Han MK, Martinez FJ, Murray S, Liu LX, Chensue SW, Polak TJ, Sonstein J, Todt JC, Ames TM, Arenberg DA, Meldrum CA, Getty C, McCloskey L, Curtis JL. Cytotoxic potential of lung CD8(+) T cells increases with chronic obstructive pulmonary disease severity and with in vitro stimulation by IL-18 or IL-15. J Immunol. 2010 Jun 1;184(11):6504-13. doi: 10.4049/jimmunol.1000006. Epub 2010 Apr 28. PMID 20427767
- [Result] Freeman CM, Martinez FJ, Han MK, Ames TM, Chensue SW, Todt JC, Arenberg DA, Meldrum CA, Getty C, McCloskey L, Curtis JL. Lung dendritic cell expression of maturation molecules increases with worsening chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2009 Dec 15;180(12):1179-88. doi: 10.1164/rccm.200904-0552OC. Epub 2009 Sep 3. PMID 19729666
- [Result] Freeman CM, Martinez CH, Todt JC, Martinez FJ, Han MK, Thompson DL, McCloskey L, Curtis JL. Acute exacerbations of chronic obstructive pulmonary disease are associated with decreased CD4+ & CD8+ T cells and increased growth & differentiation factor-15 (GDF-15) in peripheral blood. Respir Res. 2015 Aug 5;16(1):94. doi: 10.1186/s12931-015-0251-1. PMID 26243260
- See also: COPD Foundation — http://www.copdfoundation.org/
- See also: Training Grant in Lung Disease — http://www.med.umich.edu/intmed/pulmonary/edu/mtp.htm
- See also: Graduate Program in Immunology, University of Michigan — http://www.med.umich.edu/immprog/